CLINICAL TRIAL: NCT02415920
Title: The Influence of Intranasal Oxytocin on Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Frances Chen, Dr. Frances Chen, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H14-02448
Record Dates: First submitted 2015-03-31; First posted 2015-04-14 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: Investigating oxytocin's effects; human communication
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): These participants will receive 24 international units (IU) of oxytocin via a nasal spray.
  Interventions: Drug: Oxytocin
- Control - Placebo (Placebo Comparator): These participants will receive 24 international units (IU) of a saline solution via a nasal spray.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Participants will be randomly assigned to intra-nasally administer either oxytocin or a placebo on their first visit and then they will receive the other spray during their second visit.
  Other Names: Syntocinon
  Arms: Experimental
Drug: Placebo — Participants will be randomly assigned to intra-nasally administer either oxytocin or a placebo on their first visit and then they will receive the other spray during their second visit.
  Arms: Control - Placebo

SUMMARY:
This study investigates whether oxytocin, a neuropeptide known for its role in social bonding, influences the outcomes of persuasive communications and several primary evolutionary goals. Participants will be given either oxytocin or placebo on their first visit and then they will receive the other spray during their second visit. At each visit, participants will engage in several psychosocial tasks to assess the role of oxytocin on receptiveness to opposing opinions, navigating the spatial environment, mating and parenting goals. Participants' attitudes and behaviours will be compared across the different conditions.

DETAILED DESCRIPTION:
Oxytocin is a naturally occurring hormone, commonly known for its role in social approach, bonding, and trust. The present study is designed to investigate whether and how oxytocin may affect communication outcomes--specifically, by influencing trust of people presenting opinions that participants disagree with.

Healthy adult volunteers will intranasally administer 24 IU of oxytocin at one visit and placebo (saline) solution at another visit. Participants will then view photos of speakers presenting opinions on various socio-political issues which the participants disagree with. Participants will complete questions about their psychological reactions (e.g., anger, receptiveness) to the opinions presented. After reporting on their receptiveness to the opposing opinions, participants will begin the attentional tasks. In the attentional tasks, participants will be seated in front of a computer while an eyetracker records their eye movements and attentional gaze. First, participants will view two images presented simultaneously at either ends of the computer screen; each image pair will depict a a) baby and a food, b) baby and an attractive opposite sex target, or c) food and an attractive opposite sex target. Next, participants will view a series of images exclusively depicting one attractive opposite-sex target at a time; attentional bias away from faces and towards bodies (indicative of short-term mating interest; Bolmont, Cacioppo, & Cacioppo, 2014) will be tracked. After each photograph has been viewed for a fixed duration, the participant will answer a question assessing their likelihood of engaging in a one-night stand with the person pictured. After this second part of the task, we will gather saliva samples via passive drool collection. These samples will be later assayed for testosterone. Next participants will complete a measure of visual attention in which they will identify target stimuli (e.g. letters) on a computer screen via keyboard press.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult volunteers

Exclusion Criteria:

* Currently have a diagnosed mental illness or are in psychiatric or psychotherapeutic treatment.
* Are taking endocrinologically or psychoactive drugs (e.g. psychotropic drugs such as antipsychotics, antidepressants, sedatives, or sleeping pills)
* Are taking anti-hypertensive drugs or drugs with QTc prolongation
* Abuse drugs or alcohol
* Suffer from any significant medical illness, such as heart disease/cardiovascular disease, kidney disease, endocrinological disorders, or neurological disorders.
* Are not found to be physically healthy after a required prescreen questionnaire created by a doctor
* Allergic to preservatives (e.g. paragons) found in nasal sprays
* Pregnant/breastfeeding
* Are currently involved in other clinical studies in which drugs are administered.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Communication Outcomes | 60-90 minutes
  Participants will answer a series of questions regarding their reactions (e.g., anger, receptiveness) to the speakers and the opinions presented in the photos. It is expected that when participants receive oxytocin they will be more receptive to opposing opinions compared to when they receive the placebo. Participants may also have differing levels of receptiveness depending on whether the person expressing the opinion comes from their ingroup or outgroup.

SECONDARY OUTCOMES:
Appetite | 60-90 minutes
  We predict that when participants receive oxytocin they will spend less time looking at photos of food compared to when they receive the placebo.
Short vs. Long-Term mating orientation | 60-90 minutes
  When participants receive oxytocin they will spend more time looking at human infants, less time looking at attractive opposite sex others (especially the bodies of those opposite sex others; additionally, they will exhibit lower testosterone reactivity to images of attractive opposite sex targets and report weaker desires to engage in short-term romantic relationships in general.
Peripheral narrowing of attention | 60-90 minutes
  When participants receive oxytocin they will exhibit less peripheral narrowing on a computerized visual attention task compared to when they receive a placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chen, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Kenny Psychology Building, Vancouver, British Columbia, Canada